CLINICAL TRIAL: NCT01989013
Title: Effect on Parkinson's Disease After Therapeutic Induction of CranioSacral Integrated Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zia, Al Raza (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CST001
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Craniosacral therapy; cranial osteopathy
MeSH Terms: conditions — Parkinson Disease | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- biweekly intervention (Other): biweekly intervention
  Interventions: Other: biweekly intervention

INTERVENTIONS:
Other: biweekly intervention — 10 step craniosacral therapy protocol through manual therapy at feet , thoracic diaphragm, neck and cranium
  Other Names: manual therapy

SUMMARY:
We are studying & researching the effect of CranioSacral Integrative therapy on Parkinson's Diseased Patients for 3 months. With a therapeutic induction via manual CranioSacral integrative therapy for 90 minutes per session with a total of 2 session divided equally in a month (biweekly intervention). At the end of 3 months each patient will have total of 9 hours of CranioSacral Integrative therapy induced, we will document the symptoms and shortcomings of the patients at evaluation, before and after therapeutic treatment on a measured scale ranging from 1-10. Finally graphically and statistically measure the quality of change in the symptoms at the end of 3 months and provide executive summary of the research finding, which the investigators expect to be a positive one.

DETAILED DESCRIPTION:
We are studying & researching the effect of CranioSacral I therapy on Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* must be Diagnosed with Parkinson's Disease

Exclusion Criteria:

* Anyone without Parkinson's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2014-02; Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
reduction in tremors due to Parkinson's disease in the patient | 3 months
  Measurement of the tremors and quality of the coordination of the medial leminiscus system on 1-10 (1 being zero tremors and 10 being out of control tremors) scale at the evaluation and at beginning and at the end of each treatment session and in the end will provide a graphical and statistical display in the change in the tremors relative to the therapeutic induction

SECONDARY OUTCOMES:
Quality of Proprioception | 3 months
  will evaluate the patients ability to move within space and time with certain precision and measure it on a scale of 1-10 (1 being very precise with fine motor movement and 10 being out of control fine motor movements)at the time of evaluation and at the beginning and end of each therapeutic treatment and finally document it graphically and statistically, the change in the overall motor movements like walking and quality of gait.

OTHER OUTCOMES:
Overall emotional State and sleep quality | 3 months
  will evaluate the overall emotional and sleeping habits on the measurement scale of 1-10 where 1 being emotionally stable and positive with 8 hours of quality sleep and 10 being emotionally unstable and have less than 4 hours of sleep at night and at the end of research will graphically and statistically provide the outcome of the above mentioned measure.

CONTACTS AND LOCATIONS:
Overall Officials: Al Raza, CST, Principal Investigator — IBR, Inc.
Locations (1):
- Naturalmed therapy, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No